CLINICAL TRIAL: NCT00001431
Title: A Phase I Trial of Gemcitabine and Radiation in Locally Advanced Unresectable Cancer of the Pancreas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950075; 95-C-0075
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-11

CONDITIONS: Gastrointestinal Neoplasms; Pancreatic Neoplasms
Keywords: Combined Modality; GI Cancer; Pancreatic Cancer; Radiotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine

SUMMARY:
Radiotherapy plus Single-Agent Chemotherapy/Radiosensitization. Involved-field irradiation using 4-15 MV photons; plus Gemcitabine, NSC-613327.

DETAILED DESCRIPTION:
This is a Phase I trial of gemcitabine given weekly as a 30 minute infusion administered concurrently with radiation in patients with locally advanced or locally recurrent pancreatic carcinoma. Patients will be treated with external beam radiation therapy in a standard manner. Gemcitabine will be administered as a 30 minute infusion beginning on the first day of irradiation and weekly afterwards for a total of 5 doses. Patients will be assessed clinically for acute toxicity which will be graded per RTOG and DCT toxicity grading system.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically or cytologically proven unresectable adenocarcinoma of the pancreas or ampulla of Vater. Surgical consult at NCI confirming unresectability fulfills requirement.

Unresectable disease defined as tumor with: Gross involvement of regional nodes or direct extension to any of the following sites: Duodenum, Spleen, Bile duct , Colon, Peripancreatic tissue, Adjacent large vessels, Stomach.

Metastatic disease requiring local radiotherapy allowed. No CNS metastasis.

No lymphomas or neuroendocrine tumors.

No peritoneal carcinomatosis.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: More than 4 weeks since immunotherapy.

Chemotherapy:

No prior chemotherapy for newly diagnosed disease.

More than 4 weeks since chemotherapy for recurrent disease (6 weeks since nitrosoureas, mitomycin, or suramin).

Endocrine Therapy: More than 4 weeks since hormonal therapy.

Radiotherapy:

No prior radiotherapy for newly diagnosed disease.

No prior abdominal or pelvic radiotherapy.

More than 4 weeks since radiotherapy for recurrent disease. No prior radiotherapy for locally advanced disease after resection allowed.

Surgery:

Prior resection allowed.

Biliary decompression or gastric bypass allowed.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0-2.

Hematopoietic:

ANC greater than 2,000/mm(3).

Platelets greater than 100,000/mm(3).

Hepatic: AST/ALT no greater than 2.5 times normal.

Renal:

Creatinine less than 1.5 mg/dL.

Creatinine clearance at least 60 mL/min,

Cardiovascular:

No myocardial infarction within 6 months.

No unstable angina.

No congestive heart failure (NYHA class III/IV).

OTHER:

HIV seronegative.

No medical or psychiatric contraindication to protocol therapy.

No concurrent malignancy other than: Skin cancer, Cervical carcinoma in situ.

No pregnant or nursing women.

Adequate contraception required of fertile patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1995-02; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Morohoshi T, Held G, Kloppel G. Exocrine pancreatic tumours and their histological classification. A study based on 167 autopsy and 97 surgical cases. Histopathology. 1983 Sep;7(5):645-61. doi: 10.1111/j.1365-2559.1983.tb02277.x. PMID 6313514
- [Background] Rosenberg JM, Welch JP, Macaulay WP. Cancer of the head of the pancreas: an institutional review with emphasis on surgical therapy. J Surg Oncol. 1985 Mar;28(3):217-21. doi: 10.1002/jso.2930280315. PMID 2579295